CLINICAL TRIAL: NCT05849844
Title: Tympanoseal (Tympanic Membrane Device) Clinical Study
Brief Title: Tympanoseal Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grace Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022.01
Record Dates: First submitted 2023-04-13; First posted 2023-05-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tympanoseal (Experimental): All subjects will receive the Tympanoseal device that will be placed during a surgical procedure.
  Interventions: Device: Tympanoseal

INTERVENTIONS:
Device: Tympanoseal — All subjects will receive the Tympanoseal device that will be placed during a surgical procedure

SUMMARY:
The purpose of this investigational study is to assess the ability of Tympanoseal (sodium/calcium alginate), an investigational device, to act as a scaffold during healing of the tympanic membrane. Tympanoseal is intended for use following removal or extrusion of indwelling tympanostomy tubes or traumatic injury of the tympanic membrane.

DETAILED DESCRIPTION:
This study will provide data on the safety and the ability of sodium/calcium alginate gels to act as a scaffold capable of occluding a tympanic membrane perforation over the duration of complete healing. Tympanoseal could be used in cases where cartilage or fat graft tympanoplasty would be indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over 2 years of age at enrollment
2. Documentation of a retained tympanostomy tube or perforation less than 5 mm not on the edge of the tympanic membrane.
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal guardian and ability for subject to comply with the requirements of the study

Exclusion Criteria:

1. Active otorrhea or otitis media
2. Otorrhea or otitis media within 4 weeks prior to the operation
3. History of cholesteatoma
4. Perforations on the edge of the tympanic membrane
5. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
6. Subject is taking systemic/oral corticosteroids
7. Subject will require the continued use of any type of topical otic medication to the ear(s) with Tympanoseal

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with healed tympanic membrane perforations. | 12 weeks
  The purpose of this investigational study is to assess the safety of Tympanoseal when used during the healing process. Subject will be observed during the study and the the healing process of the tympanic membrane. Information will be gathered via report forms during regular visits of the patient to the investigator.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 12 weeks
  Determine if any adverse events occur during presence of material on tympanic membrane.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Michigan Ear Institute, Farmington Hills, Michigan
  - Methodist Le Bonheur, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No